CLINICAL TRIAL: NCT05279040
Title: Long-term Effects of Elexacaftor/Tezacaftor/Ivacaftor (Trikafta) on Exertional Symptoms, Exercise Performance, Ventilatory Responses, and Body Composition in Adults With Cystic Fibrosis
Brief Title: Trikafta Exercise Study in Cystic Fibrosis
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jordan Guenette, Director of Cardiopulmonary Exercise Physiology Laboratory, University of British Columbia
Other Study IDs: H21-02125
Record Dates: First submitted 2021-11-08; First posted 2022-03-15 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Cystic Fibrosis; Lung Diseases
Keywords: Dyspnea; Exercise; Trikafta
MeSH Terms: conditions — Cystic Fibrosis; Lung Diseases; Dyspnea; Motor Activity | interventions — elexacaftor, ivacaftor, tezacaftor drug combination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cystic Fibrosis Patients: Participants diagnosed with cystic fibrosis who will be initiating Trikafta treatment
  Interventions: Drug: Trikafta

INTERVENTIONS:
Drug: Trikafta — Elexacaftor/Tezacaftor/Ivacaftor combination therapy
  Other Names: Elexacaftor/Tezacaftor/Ivacaftor

SUMMARY:
Shortness of breath (dyspnea) during exercise is a major source of distress and is a commonly reported symptom in patients with cystic fibrosis (CF). A recent drug treatment option known as Trikafta, which contains elexacaftor, tezacaftor, and ivacaftor, may be used in patients with CF to help improve lung health. However, the effects of this combination therapy on dyspnea and exercise performance, a known predictor of survival in CF, are not clear. The investigators aim to understand the effects of Trikafta on these symptoms and to gain new insight into the potential health improvements in CF from using this treatment option.

DETAILED DESCRIPTION:
Justification: Advances in therapies and patient care have led to dramatic improvements in CF survival. Consequently, CF patients are living longer with varying degrees of lung function impairment. Dyspnea is a commonly reported symptom in CF that adversely impacts quality of life. Recently, elexacaftor/tezacaftor/ivacaftor (Trikafta), a combination drug therapy, was approved by Health Canada for use in CF patients. Exercise capacity is an important outcome parameter in CF and is a strong predictor of disease prognosis including survival. Although previous research in patients on elexacaftor/tezacaftor/ivacaftor combination therapy reported improved respiratory symptoms and lung function, it remains uncertain as to whether this translates into improvements in exercise performance. Stressing the respiratory system to its physiologic limits through exercise might provide a more sensitive outcome measure to evaluate the response to cystic fibrosis transmembrane regulator (CFTR) modulator therapy. Studies on another CFTR modulator therapy combining lumacaftor and ivacaftor, have shown inconclusive results on exercise tolerance in patients with CF when evaluated using an incremental work rate exercise test protocol. However, a far more clinically and physiologically relevant protocol in evaluating treatment effects is to use constant work rate exercise tests and to evaluate dyspnea at standardized submaximal exercise times. Additionally, changes in body composition shown to result from CFTR modulator therapy may also have contributed to these inconclusive findings; however, body composition has not been evaluated in previous CFTR studies.

Purpose: The purpose of this study is to determine the various factors that cause shortness of breath (or dyspnea) in patients with cystic fibrosis (CF) and to determine how treatment with Trikafta can manipulate these factors to improve shortness of breath and exercise capacity.

Hypothesis: The investigators hypothesize that Trikafta will reduce dyspnea intensity ratings and improve exercise capacity. These improvements will be associated with improvements in the ventilatory response to exercise.

Objectives: To perform detailed cardiopulmonary exercise testing before and after the initiation of Trikafta to evaluate its effect on exertional dyspnea and exercise capacity, and to evaluate potential physiological mechanisms of improvement and the impacts of changes in body composition.

Research Design: Observational study conducted over 4 visits. Participants with CF will report to the Cardiopulmonary Exercise Physiology (CPEP) Laboratory on four separate occasions. Visit 1 and 2 will occur before the participants go on drug (Trikafta) and will be separated by a minimum of 48 hours between visits. Visit 3 and 4 will occur at 12 months and 24 months after initiating drug, respectively. On visit 1, participants will complete medical history screening, anthropometric measurements, and a symptom limited incremental cycle exercise test to determine peak incremental work rate. On visit 2, participants will undergo a dual-energy X-ray absorptiometry (DEXA) scan, chronic activity-related dyspnea questionnaires, quality of life questionnaires, physical activity questionnaires, pulmonary function testing, and a constant-load cycle exercise test at 80% of peak incremental work rate. Visits 3 and 4 will include chronic activity-related dyspnea questionnaires, quality of life questionnaires, physical activity questionnaires, a DEXA scan, pulmonary function testing, and a constant-load cycle exercise test at 80% of peak incremental work rate. Data from the constant-load cycle exercise tests performed on visits 2, 3, and 4 will address our hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF and at least one copy of the F508del mutation in the cystic fibrosis transmembrane conductance regulator (CFTR) gene
* Plan to initiate Trikafta by the treating physician within 30 days of the enrolment visit
* Aged 19 years or older
* Stable clinical status based on clinical judgment of the treating physician
* Forced Expiratory Volume in 1 second (FEV1.0) < 90% predicted
* Body mass index greater than 16 or less than 30 kg/m^2
* Currently non-smoking or a past smoking history of less than 20 pack-years
* Able to read and understand English
* Fully vaccinated (at least 2 doses) for Covid-19

Exclusion Criteria:

* A disease other than CF that could importantly contribute to dyspnea or exercise limitation
* Chronic airway infection with Mycobacterium abscessus, Burkholderia cepacia complex, or other organisms with infection control implications based on the treating physicians
* Contraindications to clinical exercise testing
* Use of supplemental oxygen or desaturation less than 85% with exercise
* Diagnosis of pneumothorax in the past 4 weeks
* History of organ transplantation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The CF patients will be recruited from the St. Paul's Hospital UBC Adult CF Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Iso-time Dyspnea Rating From Baseline (Visit 2) to Visit 3 and 4 During Constant-load Exercise Tests. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Dyspnea intensity and unpleasantness ratings measured using the Borg 0-10 category ratio scale. The intensity of the sensation is how strong or how much breathing sensation the participant feels, while the unpleasantness of the sensation is how bad or how distressed it makes the participant feel. On the Borg 0-10 category ratio scale range, "0" represents no dyspnea intensity and unpleasantness (i.e., better outcome), while "10" represents the most intense or unpleasant dyspnea (i.e., worse outcome).
  Borg dyspnea intensity and unpleasantness ratings taken at iso-time, defined as the maximum time achieved on constant-load exercise tests performed on visits 2, 3, and 4 will be used in the analysis.

SECONDARY OUTCOMES:
Change From Baseline Exercise Capacity (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Endurance time measures from the start of exercise to exercise cessation on constant-load exercise tests performed on visits 2, 3, and 4 will be used in the analysis.
Change From Baseline Body Composition (Body Fat Mass) Measurements (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Standard measures of body fat mass in units of grams (g) will be performed by dual-energy X-ray absorptiometry (DEXA) scanning using a Hologic Discovery QDR 4500 (Hologic Inc., Bedford, MA.).
  DEXA scans will be performed before the initiation of Trikafta treatment (Visit 2), 12 months after drug initiation (Visit 3), and 24 months after drug initiation (Visit 4).
Change From Baseline Body Composition (Lean Body Mass) Measurements (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Standard measures of lean body mass in units of grams (g) will be performed by dual-energy X-ray absorptiometry (DEXA) scanning using a Hologic Discovery QDR 4500 (Hologic Inc., Bedford, MA.).
  DEXA scans will be performed before the initiation of Trikafta treatment (Visit 2), 12 months after drug initiation (Visit 3), and 24 months after drug initiation (Visit 4).
Change From Baseline Body Composition (Bone Mineral Content) Measurements (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Standard measures of bone mineral content in units of grams (g) will be performed by dual-energy X-ray absorptiometry (DEXA) scanning using a Hologic Discovery QDR 4500 (Hologic Inc., Bedford, MA.).
  DEXA scans will be performed before the initiation of Trikafta treatment (Visit 2), 12 months after drug initiation (Visit 3), and 24 months after drug initiation (Visit 4).
Change From Baseline Body Composition (Bone Mineral Density) Measurements (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Standard measures of bone mineral density in units of grams/centimetres^2 (g/cm^2) will be performed by dual-energy X-ray absorptiometry (DEXA) scanning using a Hologic Discovery QDR 4500 (Hologic Inc., Bedford, MA.).
  DEXA scans will be performed before the initiation of Trikafta treatment (Visit 2), 12 months after drug initiation (Visit 3), and 24 months after drug initiation (Visit 4).
Change From Baseline Body Composition (Fat Percentage) Measurements (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Standard measures of fat percentage (%) will be performed by dual-energy X-ray absorptiometry (DEXA) scanning using a Hologic Discovery QDR 4500 (Hologic Inc., Bedford, MA.).
  DEXA scans will be performed before the initiation of Trikafta treatment (Visit 2), 12 months after drug initiation (Visit 3), and 24 months after drug initiation (Visit 4).
Change From Baseline Cardiorespiratory Responses (Heart Rate) During Constant-load Exercise Tests (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Heart rate measured in units of beats per minute (beats/min)
Change From Baseline Cardiorespiratory Responses (Blood Pressure) During Constant-load Exercise Tests (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Blood pressure measured in units of millimetres of mercury (mmHg).
Change From Baseline Cardiorespiratory Responses (Arterial Oxygen Saturation) During Constant-load Exercise Tests (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Arterial oxygen saturation measured in units of %oxygen (%O2).
Change From Baseline Cardiorespiratory Responses (Minute Ventilation) During Constant-load Exercise Tests (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Minute ventilation measured in units of litres per minute (l/min).
  Data will be recorded on a breath-by-breath basis and averaged over 30-second epochs in the analysis.
Change From Baseline Cardiorespiratory Responses (Oxygen Consumption Relative to Body Weight) During Constant-load Exercise Tests (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Oxygen consumption measured in units of millilitre per kilogram per minute (ml/kg/min).
  Data will be recorded on a breath-by-breath basis and averaged over 30-second epochs in the analysis.
Change From Baseline Cardiorespiratory Responses (Oxygen Consumption) During Constant-load Exercise Tests (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Oxygen consumption measured in units of litres per minute (l/min).
  Data will be recorded on a breath-by-breath basis and averaged over 30-second epochs in the analysis.
Change From Baseline Cardiorespiratory Responses (Carbon Dioxide Production) During Constant-load Exercise Tests (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Carbon dioxide production measured in units litres per minute (l/min).
  Data will be recorded on a breath-by-breath basis and averaged over 30-second epochs in the analysis.
Change From Baseline Cardiorespiratory Responses (Ventilatory Equivalent for Oxygen) During Constant-load Exercise Tests (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Ventilatory equivalent for oxygen measured as the ratio of minute ventilation over oxygen consumption.
  Data will be recorded on a breath-by-breath basis and averaged over 30-second epochs in the analysis.
Change From Baseline Cardiorespiratory Responses (Ventilatory Equivalent for Carbon Dioxide) During Constant-load Exercise Tests (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Ventilatory equivalent for carbon dioxide measured as the ratio of minute ventilation over carbon dioxide production.
  Data will be recorded on a breath-by-breath basis and averaged over 30-second epochs in the analysis.
Change From Baseline Cardiorespiratory Responses (Tidal Volume) During Constant-load Exercise Tests (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Tidal volume measured in units of litres (l).
  Data will be recorded on a breath-by-breath basis and averaged over 30-second epochs in the analysis.
Change From Baseline Cardiorespiratory Responses (Breathing Frequency) During Constant-load Exercise Tests (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Breathing frequency measured in units of breaths per minute (breaths/min).
  Data will be recorded on a breath-by-breath basis and averaged over 30-second epochs in the analysis.
Change From Baseline Cardiorespiratory Responses (End-Inspiratory Lung Volume) During Constant-load Exercise Tests (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  End-inspiratory lung volumes measured in units of litres (l). Data will be derived from dynamic inspiratory capacity maneuvers.
Change From Baseline Cardiorespiratory Responses (End-Expiratory Lung Volume) During Constant-load Exercise Tests (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  End-expiratory lung volumes measured in units of litres (l). Data will be derived from dynamic inspiratory capacity maneuvers.
Reasons for Stopping Exercise During Constant-load Exercise Tests (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Upon exercise cessation, participants will be asked to verbalize their main reason(s) for stopping exercise (i.e., breathing discomfort, leg discomfort, combination of breathing and legs, or some other reason). Frequency data will be used in the analysis.
Qualitative Dyspnea Sensations (15-Item Questionnaire) During Constant-load Exercise Tests (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Upon exercise cessation, participants will be asked to select qualitative descriptors of breathlessness using an established 15-item questionnaire. Frequency data will be used in the analysis.
Qualitative Dyspnea Sensations (4-Item Descriptors) During Constant-load Exercise Tests (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Participants will be asked to select the most applicable dyspnea descriptor(s) after the intensity and unpleasantness ratings using the following 3 descriptors: (1) "my breathing requires more work and effort" (work and effort); (2) "I cannot get enough air in" (unsatisfied inspiration); (3) "I cannot get enough air out" (unsatisfied expiration). None to all three of the descriptors can be chosen at any one time. Multiple selections are permitted as long as they apply equally. Frequency data will be used in the analysis.
Qualitative Dyspnea Sensations (Multi-Dimensional Dyspnoea Profile) During Constant-load Exercise Tests (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Upon exercise cessation, participants will be asked to complete the multidimensional dyspnoea profile questionnaire with focus being placed on peak exercise (i.e., the last 30 seconds of loaded pedaling). Frequency data will be used in the analysis.
Leg discomfort During Constant-load Exercise Tests (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Leg discomfort ratings measured using the Borg 0-10 category ratio scale. On the Borg 0-10 category ratio scale range, "0" represents no leg discomfort (i.e., better outcome), while "10" represents the most intense leg discomfort ever experienced or could ever imagine experiencing (i.e., worse outcome).
  Leg discomfort ratings taken at iso-time, defined as the maximum time achieved on constant-load exercise tests performed on visits 2, 3, and 4, will be used in the analysis.
Change From Baseline Chronic Activity-related Dyspnea on the Modified Baseline Dyspnea Index (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Modified Baseline Dyspnea Index scoring dyspnea severity on a total score from 1 to 12 with lower scores indicating more dyspnea severity and higher scores indicating less dyspnea severity.
Chronic Activity-related Dyspnea on the Transition Dyspnea Index at 12 and 24 Months After Initiating Full Dose of Trikafta. | 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Transition Dyspnea Index will grade change in dyspnea intensity related to functional impairment, magnitude of task, and magnitude of effort on a scale from +3 (i.e., major improvement) to zero (i.e., no change) to -3 (i.e., major deterioration).
Change From Baseline Chronic Activity-related Dyspnea on the MMRC Scale (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Modified Medical Research Council Dyspnea Scale will grade dyspnea severity on a scale of 0 = NOT TROUBLED WITH BREATHLESSNESS EXCEPT WITH STRENUOUS EXERCISE; 1 = TROUBLED BY SHORTNESS OF BREATH WHEN HURRYING ON THE LEVEL OR WALKING UP A SLIGHT HILL; 2 = WALKS SLOWER THAN PEOPLE OF THE SAME AGE ON THE LEVEL BECAUSE OF BREATHLESSNESS OR HAS TO STOP FOR BREATH WHEN WALKING AT OWN PACE ON THE LEVEL; 3 = STOPS FOR BREATH AFTER WALKING ABOUT 100 YARDS OR AFTER A FEW MINUTES ON THE LEVEL; or 4 = TOO BREATHLESS TO LEAVE THE HOUSE OR BREATHLESS WHEN DRESSING OR UNDRESSING
Change From Baseline Chronic Activity-related Dyspnea on the Oxygen Cost Diagram (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Oxygen Cost Diagram will grade dyspnea severity by marking a point along a vertical line with lists of tasks/activities on either side of the line to indicate activities beyond the point that make the subject breathless. The distance of the point from the bottom of the line (in centimetres) will be used in the analyses.
Change From Baseline Quality of Life (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Quality of life measured using the St. George's Respiratory Questionnaire. The questionnaire is scored from 0 to 100 where higher scores indicate greater limitations.
Change From Baseline Physical Activity (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Physical activity measured in metabolic equivalents (MET)-min/week using the International Physical Activity Questionnaire (Long Form).
Change From Baseline Spirometry Measures (FEV1) (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Spirometry-derived measures of Forced Expiratory Volume in 1 second (FEV1) measured in litres (l) using a commercially available cardiopulmonary testing system (V62J Autobox, Carefusion, Yorba Linda, CA.).
Change From Baseline Spirometry Measures (FVC) (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Spirometry-derived measures of Forced Vital Capacity (FVC) measured in litres (l) using a commercially available cardiopulmonary testing system (V62J Autobox, Carefusion, Yorba Linda, CA.).
Change From Baseline Plethysmography Measures (TLC) (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Plethysmography-derived measures of Total Lung Capacity (TLC) measured in litres (l) using a commercially available cardiopulmonary testing system (V62J Autobox, Carefusion, Yorba Linda, CA.).
Change From Baseline Plethysmography Measures (VC) (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Plethysmography-derived measures of Vital Capacity (VC) measured in litres (l) using a commercially available cardiopulmonary testing system (V62J Autobox, Carefusion, Yorba Linda, CA.).
Change From Baseline Plethysmography Measures (IC) (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Plethysmography-derived measures of Inspiratory Capacity (IC) measured in litres (l) using a commercially available cardiopulmonary testing system (V62J Autobox, Carefusion, Yorba Linda, CA.).
Change From Baseline Plethysmography Measures (FRC PL) (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Plethysmography-derived measures of Functional Residual Capacity (FRC PL) measured in litres (l) using a commercially available cardiopulmonary testing system (V62J Autobox, Carefusion, Yorba Linda, CA.).
Change From Baseline Plethysmography Measures (RV) (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Plethysmography-derived measures of Residual Volume (RV) measured in litres (l) using a commercially available cardiopulmonary testing system (V62J Autobox, Carefusion, Yorba Linda, CA.).
Change From Baseline Plethysmography Measures (sRaw) (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Plethysmography-derived measures of specific airway resistance (sRaw) measured in centimetres of water per litres per seconds per litre (cmH2O/L/s/L) using a commercially available cardiopulmonary testing system (V62J Autobox, Carefusion, Yorba Linda, CA.).
Change From Baseline Pulmonary Function Measures (MVV) (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Maximal Voluntary Ventilation (MVV) measured in litres per minutes (l/min) using a commercially available cardiopulmonary testing system (V62J Autobox, Carefusion, Yorba Linda, CA.).
Change From Baseline Pulmonary Function Measures (DLCO) (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Diffusing capacity of the lungs for carbon monoxide measured in millilitres per millimetres mercury per minute (mL/mmHg/min) using a commercially available cardiopulmonary testing system (V62J Autobox, Carefusion, Yorba Linda, CA.).
Change From Baseline Pulmonary Function Measures (MIP) (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Maximum inspiratory pressure (MIP) measured in centimetres of water (cmH2O) using a commercially available cardiopulmonary testing system (V62J Autobox, Carefusion, Yorba Linda, CA.).
Change From Baseline Pulmonary Function Measures (MEP) (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Maximum expiratory pressure (MEP) measured in centimetres of water (cmH2O) using a commercially available cardiopulmonary testing system (V62J Autobox, Carefusion, Yorba Linda, CA.).
Change From Baseline Impulse Oscillometry Measures of Resistance at 5 Hz (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Impulse oscillometry derived measures of Resistance at 5 hertz (Hz) in units of centimetre of water per litre per second (cmH2O/l/sec) using a commercially available cardiopulmonary testing system (V62J Autobox, Carefusion, Yorba Linda, CA.).
Change From Baseline Impulse Oscillometry Measures of Resistance at 20 Hz (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Impulse oscillometry derived measures of Resistance at 20 hertz (Hz) in units of centimetre of water per litre per second (cmH2O/l/sec) using a commercially available cardiopulmonary testing system (V62J Autobox, Carefusion, Yorba Linda, CA.).
Change From Baseline Impulse Oscillometry Measures of Reactance (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Impulse oscillometry derived measures of Reactance in units of centimetre of water per litre per second (cmH2O/l/sec) using a commercially available cardiopulmonary testing system (V62J Autobox, Carefusion, Yorba Linda, CA.).
Change From Baseline Impulse Oscillometry Measures of Area of Reactance (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Impulse oscillometry derived measures of Area of Reactance in units of centimetre of water per litre (cmH2O/l) using a commercially available cardiopulmonary testing system (V62J Autobox, Carefusion, Yorba Linda, CA.).
Change From Baseline Impulse Oscillometry Measures of Differential Change in Resistance (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Impulse oscillometry derived measures of Differential Change in Resistance (R5-R20) expressed as a percentage (%) using a commercially available cardiopulmonary testing system (V62J Autobox, Carefusion, Yorba Linda, CA.).
Change From Baseline Sweat Chloride Levels (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Cystic fibrosis transmembrane conductance regulator (CFTR) modulating effect determined by measuring sweat chloride levels in units of mmol/L during a sweat test.
Change From Baseline Computed Tomography Phenotyping (Bronchiectasis) (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Extent of bronchiectasis scored on a range from 0 to 12 (where higher scores indicate greater extent of bronchiectasis) measured using chest computed tomography (CT) scans.
Change From Baseline Computed Tomography Phenotyping (Mucus Plugging) (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Extent of mucus plugging scored on a range from 0 to 6 (where higher scores indicate greater extent of mucus plugging) measured using chest computed tomography (CT) scans.
Change From Baseline Computed Tomography Phenotyping (Air Trapping) (Prior to Trikafta Initiation to Full Dose) at 12 and 24 Months After Initiating Full Dose of Trikafta. | Baseline (i.e., Visit 2), 12 months post Trikafta initiation (i.e., Visit 3), and 24 months post Trikafta initiation (i.e., Visit 4)
  Extent of air trapping scored on a range from 0 to 4.5 (where higher scores indicate greater extent of air trapping) measured using chest computed tomography (CT) scans.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan A Guenette, PhD, Principal Investigator — University of British Columbia
Locations (1):
- UBC Centre for Heart Lung Innovation, St. Paul's Hospital, Vancouver, British Columbia, Canada